CLINICAL TRIAL: NCT00557284
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy of Montelukast (Singulair) in Participants Ages 1 - 8 Years Diagnosed With Atopic Dermatitis Induced by Food Allergens
Brief Title: Efficacy Study of Montelukast in Atopic Dermatitis Induced by Food Allergens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: 1st Allergy & Clinical Research Center (Other)
Responsible Party: Principal Investigator, Isaac Melamed, Principle Investigator, 1st Allergy & Clinical Research Center
Organization: IMMUNOe Research Centers (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 32032
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2014-12-09 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis (Eczema) associated with food allergies
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Montelukast
  Interventions: Drug: Montelukast
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — 4 mg oral granules for ages 12 - 23 months; 4 mg chewable tablet for 2 - 5 years of age; or 5 mg chewable tablet for 6 - 8 years of of age
  Arms: 1
Drug: Placebo — Oral granules or chewable tablet, PO QD (given oral daily)
  Arms: 2

SUMMARY:
AD is a disease found in children; the focus of the study is the mechanisms associated in children with AD induced by food allergies.

This study will be a randomized, double-blind, placebo-controlled, parallel group trial conducted in participants diagnosed with atopic dermatitis and food allergies. The study duration for participants will be approximately 9 weeks. A total of 20 participants will be recruited for the entire study. Each arm will consist of 10 participants.The study will enroll 20 children, male or female, 1 - 8 years of age with atopic dermatitis (AD) associated with food allergens, previously documented by skin or RAST test, before enrollment. Atopic dermatitis and gastrointestinal (GI) symptoms will be scored and followed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate atopic dermatitis involving greater than or equal to 5% of body surface
2. Total severity score of 2 or greater for any 3 of the 4 signs and symptoms calculated by study doctor (erythema, papulation, or lichenification)
3. Positive skin or (radioallergosorbent) RAST tests by ImmunoCap to food or environmental allergens
4. GI symptoms total score of 2 by caregiver on GSRS scale revised for pediatrics

Exclusion Criteria:

1. Participants with intolerance or allergy to montelukast.
2. History of anaphylaxis requiring hospitalization.
3. No underlying renal or liver disease.
4. Participants with a diagnosis of severe asthma.
5. Participants diagnosed with primary immune deficiency.
6. Participants using sublingual immunotherapy.
7. Immunotherapy must be a maintenance dose for a minimum of 30 days.
8. If on gastrointestinal medication, 30 day stable dose before visit 1 and maintained throughout the study.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isaac R Melamed, MD, Principal Investigator — 1st Allergy & Clinical Research Center
Locations (2):
- United States (2):
  - 1st Allergy & Clinical Research Centers, Centennial, Colorado
  - 1st Allergy & Clinical Research Centers, Thornton, Colorado

REFERENCES:
- See also: Research website — http://www.immunoeresearch.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 outpatient clinics in the Denver, Colorado, metropolitan area between February 2008 and March 2009. Individual subject participation lasted for approximately 9 weeks.
Pre-assignment Details: Thirty-three subjects were screened for the trial; 20 subjects met all inclusion and exclusion criteria; 13 failed to meet all inclusion criteria.
Groups:
- Treatment Arm: Montelukast : 4 mg oral granules for ages 12 - 23 months; 4 mg chewable tablet for 2 - 5 years of age; or 5 mg chewable tablet for 6 - 8 years of of age
- Placebo Arm: Placebo : Oral granules or chewable tablet, POQD
Period: Overall Study
Arm/Group | Treatment Arm | Placebo Arm
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Placebo Arm | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 11 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (2.3) | 5.6 (1.7) | 5.5 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20
Percentage of Body Involvement [Mean (Standard Deviation); unit: percentage] — Percentage of body surface as calculated by investigator. Measurement is mean for all subjects in each arm.
  percentage | 21.67 (8.9) | 20.05 (8.1) | 20.86 (8.5)
Investigator Global Assessment (IGA) [Mean (Standard Deviation); unit: Scores on a scale] — The IGA is a six-point measure of disease severity are evaluated by the study doctor based on the overall assessment of skin lesions: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5= very severe. Measurement is the mean for all subjects in each arm.
  Scores on a scale | 2.11 (0.33) | 2.30 (0.48) | 2.20 (0.40)
PADC (caregivers assessment of disease control) [Mean (Standard Deviation); unit: Scores on a scale] — Caregiver's evaluation of disease control over the previous 7 days and will consist of a four-point scale ranging from complete control (0) to uncontrolled disease (3). Measurement is the mean for all subjects in each arm.
  Scores on a scale | 1.78 (0.67) | 1.80 (0.92) | 1.79 (0.80)
Pruritus score [Mean (Standard Deviation); unit: units on a scale] — Pruritus assessments ("itch") will be recorded for the previous 24 hours using a 4 point-scale, ranging from none (0) to severe (3). Measurement is mean of all subjects in each arm.
  units on a scale | 1.60 (0.79) | 1.17 (0.72) | 1.36 (0.30)
IL-13 [Mean (Standard Deviation); unit: pg/ml] — Serum interleukin 13 levels. Measurement is the mean for all subjects in each arm.
  pg/ml | 33.67 (30.20) | 34.70 (37.0) | 34.18 (33.60)
TNF alpha [Mean (Standard Deviation); unit: pg/ml] — Serum Tumor Necrosis Factor levels. Measurement is the mean for all subjects in each arm.
  pg/ml | 1.87 (0.87) | 5.70 (11.03) | 3.78 (5.95)
NGF [Mean (Standard Deviation); unit: pg/ml] — Serum Nerve Growth Factor levels. Measurement is the mean for all subjects in each arm.
  pg/ml | 99.78 (167.38) | 108.70 (192.35) | 104.24 (179.86)
Urine LTE4 [Mean (Standard Deviation); unit: pg/ml] — Urine Cysteinyl leukotriene 4 levels. Measurement is the mean for all subjects in each arm.
  pg/ml | 52.90 (40.20) | 66.65 (62.90) | 59.77 (51.55)
IgE [Mean (Standard Deviation); unit: kU/L] — Serum Immunoglobulin E levels. Measurement is the mean for all subjects in each arm.
  kU/L | 432.20 (887.90) | 392.40 (441.00) | 412.30 (664.45)
GSRS [Mean (Standard Deviation); unit: Scores on a scale] — GI symptoms will be recorded weekly on *GSRS validated scale adjusted for pediatrics (*Gastrointestinal Symptoms in Patients with Irritable Bowel Syndrome and Peptic Ulcer Disease). This scale measures 7 different GI symptoms (1. abdominal pain; 2. nausea and vomiting; 3. abdominal dissention; 4. decreased passage of stools; 5. increased passage of stools; 6. loose stools; 7. hard stools) with severity ranges from 0 - 3 (maximum total of 21 - most severe). Measurement is the mean for all subjects in each arm.
  Scores on a scale | 4.67 (2.5) | 5.0 (2.4) | 4.83 (2.45)

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change in Serum and Urinary Inflammatory Marker Levels
Description: Mean change in levels from baseline to study visit 4 (week 1 compared to week 9)for interleukin 3 (IL3), tumor necrosis factor alpha (TNF alpha), nerve growth factor (NGF), and urinary leukotriene E4 (LTE4)
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 9 | 11
pg/ml
  IL3 | -9.0 (43.9) | -7.9 (53.7)
  TNF alpha | 2.3 (5.5) | -16.4 (13.6)
  NGF | 30.9 (306.7) | -58.8 (198.3)
  Urine LTE4 | -2.1 (46.2) | -20.42 (65.0)

2. Secondary Outcome: Mean Change in Serum IgE Levels
Description: Mean change in serum levels of IgE from baseline to study visit 4 (week 1 compared to week 9) for all subjects in each arm.
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: kU/L
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 9 | 11
kU/L | 100.5 (355.6) | 216.1 (505.9)

3. Primary Outcome: Change in Percentage of Body Involvement
Description: Change in percentage of body involvement from baseline to study visit 4 (week 1 compared to week 9) for all subjects in each arm for AD as measured by study investigator
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: Change of percentage in body involvement
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 9 | 11
Change of percentage in body involvement | -2.0 (12.2) | 0.15 (20.2)

4. Primary Outcome: Mean Change in Investigator Global Assessment (IGA)
Description: The mean change in IGA from baseline to study visit 4 (week 1 compared to week 9) for all subjects in each arm. The IGA is a six-point measure of disease severity and is evaluated by the investigator based on the overall assessment of skin lesions: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5= very severe.
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 9 | 11
units on a scale | -.11 (1.7) | -.70 (.95)

5. Primary Outcome: Mean Change in PADC (Caregivers Perception of Disease Control)
Description: Mean change in PADC from baseline to study visit 4 (week 1 compared to week 9) for all subjects in each arm. Caregiver's evaluation of disease control over the previous 7 days and will consist of a four-point scale ranging from complete control (0) to uncontrolled disease (3)
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 9 | 11
units on a scale | -.78 (1.1) | -0.10 (1.4)

6. Primary Outcome: Mean Change in Pruritus
Description: Mean change in pruritus scores from baseline to study visit 4 (week 1 compared to week 9) for all subjects in each arm. Pruritus assessments ("itch") will be recorded for the previous 24 hours using a 4 point-scale, ranging from none (0) to severe (3). Scores are cumulative per week.
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 9 | 11
units on a scale | -0.82 (0.78) | 0.32 (0.45)

7. Primary Outcome: Mean Change in Weekly Use of Rescue Medication for AD Flare-up - Cetirizine and/or 10% Hydrocortisone Cream
Description: Average of weekly use of cetirizine and/or 10% hydrocortisone cream will be compared for all subjects in each arm from week 1 to week 9. Flare-up is defined as a worsening of the disease that is unacceptable to the participants and leads to second line topical steroid use and/or liquid anti-histamine use. Measurement is noted as 1 for daily use (does not correspond to multiple uses per day).
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 9 | 11
days/week
  Cetirizine use | -0.56 (0.88) | 0.91 (2.1)
  10% Hydrocortisone cream use | 0.78 (2.7) | 2.0 (3.3)

8. Secondary Outcome: Mean Change in (Gastrointestinal Symptom Rating Scale) GSRS
Description: The mean change from baseline to study visit 4 (week 1 compared to week 9) in GRGS scores (GI symptoms will be recorded on *GSRS validated scale adjusted for pediatrics (*Gastrointestinal Symptoms in Patients with Irritable Bowel Syndrome and Peptic Ulcer Disease) for all subjects in each arm.This scale measures 7 different GI symptoms (1. abdominal pain; 2. nausea and vomiting; 3. abdominal dissention; 4. decreased passage of stools; 5. increased passage of stools; 6. loose stools; 7. hard stools) with severity ranges from 0 - 3 for each point (0 being no complaint and 3 being most severe for a maximum total of 21).
Time Frame: Baseline and 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 9 | 11
units on a scale | -3.03 (3.1) | -4.1 (3.1)

ADVERSE EVENTS:
Arm/Group | Treatment Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No